CLINICAL TRIAL: NCT02417389
Title: Efficacy of a Calcimimetic (Cinacalcet) in the Long Term Control of Patients With Primary Hyperparathyroidism
Brief Title: Efficacy of Cinacalcet in the Control of Primary Hyperparathyroidism
Acronym: CA-PHP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Maria Luisa Bianchi, M.D., Istituto Auxologico Italiano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02A605_2006
Record Dates: First submitted 2015-04-08; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Hyperparathyroidism, Primary; Osteoporosis
Keywords: primary hyperparathyroidism; hypercalcemia; osteoporosis; bone turnover; bone mineral density; fractures
MeSH Terms: conditions — Hyperparathyroidism, Primary; Osteoporosis; Hypercalcemia; Fractures, Bone | interventions — Cinacalcet; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cinacalcet (Experimental): Phase 1 (12 months): all patients treated with cinacalcet alone; Phase 2 (12 months): all patients treated with cinacalcet plus alendronate
  Interventions: Drug: cinacalcet; Drug: Alendronate

INTERVENTIONS:
Drug: cinacalcet — During Phase 1 (months 1-12): oral administration; 30 mg twice/day (dose to be increased if needed).
  Other Names: Mimpara
Drug: Alendronate — During Phase 2 (months 13-24): oral administration; 70 mg once/week (in addition to cinacalcet 30 mg twice/day as during Phase 1).
  Other Names: Alendronic acid; Fosamax

SUMMARY:
To assess the efficacy and safety of treatment with cinacalcet and with cinacalcet plus alendronate in controlling bone loss induced by primary hyperparathyroidism.

DETAILED DESCRIPTION:
The project was conducted at the Istituto Auxologico Italiano, IRCCS, Milano (Italy).

Principal Investigator: Maria Luisa Bianchi, M.D., Nephrologist, Bone Metabolism Unit, Istituto Auxologico Italiano IRCCS, Milan, Italy

Other investigators:

Silvia Vai, M.D., endocrinologist, Bone Metabolism Unit, Istituto Auxologico Italiano IRCCS, Milan, Italy Francesca Broggi, Dr., biologist, Bone Metabolism Unit, Istituto Auxologico Italiano IRCCS, Milan, Italy Luca Persani, M.D., Endocrinologist, University of Milan & Division of Endocrine and Metabolic Diseases, Istituto Auxologico Italiano IRCCS, Milan, Italy

Introduction Cinacalcet is an orally active second-generation calcimimetic drug. Cinacalcet increases the sensitivity of calcium receptors located on the surface of parathyroid cells, thus inhibiting parathyroid hormone (PTH) secretion (which is increased in hyperparathyroidism). Cinacalcet has been approved by FDA and EMEA for the use in dialyzed patients affected by chronic renal failure with uncontrolled secondary hyperparathyroidism, on the basis of three 6-month double-blind placebo-controlled studies on more than 1,100 patients.

PTH secretion and parathyroid cell proliferation are regulated by the serum levels of ionized calcium (Ca++). The mechanism is based on the binding of the Ca++ ion to a G-protein coupled membrane receptor (GPCR), called Calcium Sensing Receptor (CaR). With low circulating levels of Ca++ or with an alteration of the calcium-receptor binding, higher amounts of PTH are secreted, hyperparathyroidism develops, and in the long term systemic alterations (bone mineral density (BMD) reduction, increased fracture risk, hypercalciuria, renal stones, hypertension, etc.) appear.

Substances with calcimimetic action, such as Cinacalcet, have been recently developed. Until now, Cinacalcet has been mainly used in hyperparathyroidism secondary to renal insufficiency.

In this condition, Cinacalcet has been proven effective in reducing the circulating PTH to acceptable levels, obtaining the normalization of serum Ca++ and phosphate levels in about 50% of cases. Moreover, the drug is usually well tolerated. Side effects (essentially nausea and vomiting) are reported in about 30% of cases.

Pilot studies have confirmed the efficacy of Cinacalcet in maintaining a normal calcemia in the long term also in patients with primary hyperparathyroidism (PHP) due to adenoma or carcinoma of one parathyroid gland.

For this reason, the investigators proposed to use of Cinacalcet in cases of PHP, in which surgical intervention was not possible, and its use in combination with oral alendronate in the presence of osteopenia/osteoporosis.

Study objectives

* To assess the efficacy and safety of long-term Cinacalcet treatment in patients with PHP, who are not operable, or in whom the localization of the parathyroid adenoma has not been possible.
* To assess the efficacy of a combined therapy with Cinacalcet and alendronate in controlling the bone loss induced by PHP.

Study design: prospective, single-arm, 24-month study, organized in two phases. During Phase 1, all patients were treated with Cinacalcet alone for 12 months. During Phase 2, all patients were treated with Cinacalcet (as before) plus oral alendronate (70 mg once weekly) for another 12 months.

The study was conducted in accordance with the Good Clinical Practice (GCP) rules, and was approved by the Ethical Committee of the Istituto Auxologico Italiano, IRCCS.

Timelines

The study was organized as follows:

* 10 months for patient enrolment
* 24 months for the study (Phase 1 plus Phase 2)
* 6 months for the analysis of results

The enrolment was started after the approval of the protocol and the commitment of the manufacturing Company to supply the Cinacalcet.

Study population 22 patients with PHP, who are not operable, or in whom the localization of the parathyroid adenoma has not been possible, and with reduced bone density (T-score ≤ -2 at spine or hip) were included in the study. All patients were post-menopausal women.

Patients were included in the study, according to the pre-defined inclusion criteria (all 5 criteria must be met) and exclusion criteria (none of these criteria must be met).

Definition of PHP: serum intact PTH level higher than 65 ng/ml on at least two determinations during the 12 months before the start of the study (after exclusion of severe hypovitaminosis D), and serum calcium higher than 10.4 mg/dl.

All patients were studied in advance with parathyroid ecography or neck CT, and scintigraphy with Sestamibi.

At the time of enrolment, the following exams were done:

1. evaluation of phosphate and calcium metabolism (blood: intact parathyroid hormone, total calcium, ionized calcium, phosphate, creatinine, 25-hydroxy-vitamin D 1,25-dihydroxy-vitamin D, bone-specific alkaline phosphatase, C-terminal telopeptide; urine: calciuria 24-hours, phosphaturia 24-hours, N-terminal telopeptide, creatinine clearance)
2. bone density evaluation (DXA scan: radius, lumbar spine, proximal femur, and total body)
3. general evaluation (liver function, blood cell count, renal function (serum creatinine and creatinine clearance)

Treatment and follow-up The initial treatment regimen was 30 mg of Cinacalcet twice a day, at 12-hour intervals.

The follow-up was done as follows:

* 2 weeks after starting Cinacalcet, the plasma levels of total calcium and intact PTH were measured. If the calcemia was still above 10.6 mg/dl, the Cinacalcet dose was doubled (60 mg twice a day).
* 4 weeks after starting Cinacalcet, the following biochemical parameters were measured: blood: PTH, total calcium, ionized calcium, phosphate, creatinine, liver function, blood cell count; urine: calciuria 24-hours, phosphaturia 24-hours, N-terminal telopeptide, creatinine clearance. If calcemia was still above 10.6 mg/dl, the Cinacalcet dose was increased 90 mg twice a day.
* every 8 weeks, the following biochemical parameters were measured: blood: PTH, calcium, ionized calcium, phosphate, creatinine, liver function, blood cell count; urine: calciuria 24-hours, phosphaturia 24-hours, N-terminal telopeptide, creatinine clearance.
* after 12 months of Cinacalcet therapy, the DXA scan was repeated, and oral alendronate at the dose of 70 mg weekly will be added
* at the end of the 24th month of therapy, all the exams done at the time of enrolment were repeated During the study, if serum total calcium levels decreased below 8.4 mg/dl, the Cinacalcet daily dose was halved. If serum total calcium levels were still below 8.4 mg/dl with the minimum dose of Cinacalcet (30 mg once a day), Cinacalcet was stopped.

In these cases, serum calcemia was measured again at 1-week intervals, and the Cinacalcet treatment was resumed accordingly.

All the patients' data were collected in a specially designed CRF (case report form).

Side effects and adverse reactions were appropriately recorded in the CRF. The severity of the side effects or adverse reactions were evaluated in order to decide whether the involved drug(s) should be stopped.

Adverse events (AE) were recorded in a dedicated section of the CRF, in accordance with the standard rules of clinical trials. The adverse events were classified, as usual, as serious AE (SAE) or non-serious AE (AE). For each AE severity and causality were recorded. SAEs were immediately reported to the drug manufacturer (Amgen). Appropriate clinical decisions (immediate and follow-up) were made.

According to the available literature, side effects of Cinacalcet were generally mild.

In case of severe side effects or SAE, treatment was to be stopped.

Methods All DXA scans and laboratory tests were performed at the Istituto Auxologico Italiano IRCCS.

Bone mass was measured with a dual X-ray (DXA) Hologic Discovery densitometer at distal radius, lumbar spine, hip and on total body.

Serum and urinary calcium and phosphorus were measured with standard methods. Serum bone alkaline phosphatase (BSAP) were measured by EIA (enzyme-linked immunosorbent assay; Quidel, San Diego, USA); serum C-terminal telopeptide (CTx) by immunoluminescent method (Roche Diagnostic, Monza, Italy); urinary N-terminal telopeptide of procollagen type I (NTx) by EIA (enzyme-linked immunosorbent assay; Ostex Intern. Inc., Seattle, USA). Serum intact parathyroid hormone (PTH) was measured by immunoluminescent method (Roche Diagnostic, Monza, Italy); 25-hydroxyvitamin D (25-OH D) by RIA (radioimmunological assay, DiaSorin Inc, Stillwater, USA); 1,25-dihydroxyvitamin D (1,25(OH)2 D) by radio receptor assay (Nichols Institute Diagnostics, San Juan Capistrano, USA).

Statistical methods

To evaluate the sample size, the following points were considered:

1. The study was focused on a well-characterized, homogeneous group of patients affected by PHP without the possibility of surgical removal of the adenoma, and also affected by osteopenia/osteoporosis.
2. These patients had already been followed at our Center for several years, so the risk of drop-out re was very low (estimated 10%).
3. Considering the characteristics of the study (single-arm), a confidence level of 95%, a 5% significance, a drop-out rate of 10%, the 2.5% change in BMD, a sample size of 16 patients was calculated.

On the basis of the patients coming to our attention, the investigators estimated to be able to enroll 20 patients meeting the inclusion criteria.

Data were expressed as the mean plus or minus SD. All the variables were analyzed to evaluate their normality (Shapiro-Wilk test), in order to choose the appropriate statistical tests.

To estimate the comparison of the means, after evaluating the validity assumptions, the Student's t test and one-way ANOVA were used.

Statistical significance was defined as p<0.05, two-sided. At the end of the study, the occurrence of adverse events was analyzed with descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. patients affected by moderate to severe PHP without instrumental (echography, neck CT, scintigraphy with Sestamibi) evidence of parathyroid adenoma or hyperplasia; OR patients affected by PHP and previously surgically treated, but recidivating without instrumental evidence of parathyroid adenoma or hyperplasia; OR patients affected by PHP and judged inoperable because of other pathologies
2. patients with serum total calcium between 10.5 and 12.5 mg/dl (inclusive)
3. males: age ≥50 years; females: age ≥50 years, in menopause for at least 2 years;
4. patients with reduction of bone density (T-score ≤ -2 at spine OR hip, by DXA scan)
5. informed consent signed at enrolment

Exclusion Criteria:

1. lack of informed consent;
2. presence of other diseases known to cause hypercalcemia (e.g. familial benign hypercalcemia);
3. previous or ongoing therapies interfering with calcium and bone metabolism;
4. impaired liver and/or renal function (i.e. serum aspartate aminotransferase, alanine aminotransferase and total bilirubin twice the upper limit of normal or more; creatinine clearance lower than 60 ml/min);
5. history of seizures, malignancy, myocardial infarction;
6. previous exposure to cinacalcet.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
percentage of patients reaching normal serum levels of calcium and maintaining these levels at end of Phase 1 and Phase 2. | 24 months
  calcemia measurement
percentage of patients obtaining a reduction of serum levels of calcium of at least 0.5 mg/dl below their baseline values and maintaining such reduction at end of Phase 1 and Phase 2. | 24 months
  calcemia measurement
percentage of patients obtaining an increase of spine or femoral BMD of 2.5% or more with respect to their baseline values at end of Phase 1 and Phase 2. | 24 months
  DXA BMD measurement at spine and hip

SECONDARY OUTCOMES:
reduction of serum BSAP with respect to baseline value | 12 months and 24 months
  BSAP measurement
reduction of serum CTx with respect to baseline value | 12 months and 24 months
  CTx measurement
reduction of urinary NTx with respect to baseline value | 12 months and 24 months
  NTx measurement
change of spine and femoral BMD with respect to baseline values | 12 months and 24 months
  DXA BMD measurement at spine and hip

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa BIANCHI, M.D., Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy

REFERENCES:
- [Background] Dong BJ. Cinacalcet: An oral calcimimetic agent for the management of hyperparathyroidism. Clin Ther. 2005 Nov;27(11):1725-51. doi: 10.1016/j.clinthera.2005.11.015. PMID 16368445
- [Background] Block GA, Martin KJ, de Francisco AL, Turner SA, Avram MM, Suranyi MG, Hercz G, Cunningham J, Abu-Alfa AK, Messa P, Coyne DW, Locatelli F, Cohen RM, Evenepoel P, Moe SM, Fournier A, Braun J, McCary LC, Zani VJ, Olson KA, Drueke TB, Goodman WG. Cinacalcet for secondary hyperparathyroidism in patients receiving hemodialysis. N Engl J Med. 2004 Apr 8;350(15):1516-25. doi: 10.1056/NEJMoa031633. PMID 15071126
- [Background] Lindberg JS, Culleton B, Wong G, Borah MF, Clark RV, Shapiro WB, Roger SD, Husserl FE, Klassen PS, Guo MD, Albizem MB, Coburn JW. Cinacalcet HCl, an oral calcimimetic agent for the treatment of secondary hyperparathyroidism in hemodialysis and peritoneal dialysis: a randomized, double-blind, multicenter study. J Am Soc Nephrol. 2005 Mar;16(3):800-7. doi: 10.1681/ASN.2004060512. Epub 2005 Feb 2. PMID 15689407
- [Background] Moe SM, Cunningham J, Bommer J, Adler S, Rosansky SJ, Urena-Torres P, Albizem MB, Guo MD, Zani VJ, Goodman WG, Sprague SM. Long-term treatment of secondary hyperparathyroidism with the calcimimetic cinacalcet HCl. Nephrol Dial Transplant. 2005 Oct;20(10):2186-93. doi: 10.1093/ndt/gfh966. Epub 2005 Jul 19. PMID 16030053
- [Background] Cunningham J, Danese M, Olson K, Klassen P, Chertow GM. Effects of the calcimimetic cinacalcet HCl on cardiovascular disease, fracture, and health-related quality of life in secondary hyperparathyroidism. Kidney Int. 2005 Oct;68(4):1793-800. doi: 10.1111/j.1523-1755.2005.00596.x. PMID 16164656
- [Background] Barman Balfour JA, Scott LJ. Cinacalcet hydrochloride. Drugs. 2005;65(2):271-81. doi: 10.2165/00003495-200565020-00007. PMID 15631545
- [Background] Shoback DM, Bilezikian JP, Turner SA, McCary LC, Guo MD, Peacock M. The calcimimetic cinacalcet normalizes serum calcium in subjects with primary hyperparathyroidism. J Clin Endocrinol Metab. 2003 Dec;88(12):5644-9. doi: 10.1210/jc.2002-021597. PMID 14671147
- [Background] Peacock M, Bilezikian JP, Klassen PS, Guo MD, Turner SA, Shoback D. Cinacalcet hydrochloride maintains long-term normocalcemia in patients with primary hyperparathyroidism. J Clin Endocrinol Metab. 2005 Jan;90(1):135-41. doi: 10.1210/jc.2004-0842. Epub 2004 Nov 2. PMID 15522938
- [Background] Silverberg SJ, Bilezikian JP. The diagnosis and management of asymptomatic primary hyperparathyroidism. Nat Clin Pract Endocrinol Metab. 2006 Sep;2(9):494-503. doi: 10.1038/ncpendmet0265. PMID 16957763
- [Background] Bilezikian JP, Brandi ML, Rubin M, Silverberg SJ. Primary hyperparathyroidism: new concepts in clinical, densitometric and biochemical features. J Intern Med. 2005 Jan;257(1):6-17. doi: 10.1111/j.1365-2796.2004.01422.x. PMID 15606372
- [Background] Bilezikian JP, Potts JT Jr, Fuleihan Gel-H, Kleerekoper M, Neer R, Peacock M, Rastad J, Silverberg SJ, Udelsman R, Wells SA. Summary statement from a workshop on asymptomatic primary hyperparathyroidism: a perspective for the 21st century. J Clin Endocrinol Metab. 2002 Dec;87(12):5353-61. doi: 10.1210/jc.2002-021370. No abstract available. PMID 12466320
- [Background] Jorde R, Bonaa KH, Sundsfjord J. Primary hyperparathyroidism detected in a health screening. The Tromso study. J Clin Epidemiol. 2000 Nov;53(11):1164-9. doi: 10.1016/s0895-4356(00)00239-0. PMID 11106891